CLINICAL TRIAL: NCT00003163
Title: Myeloblative Therapy With Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Myeloma and B-Cell Malignancies
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma or Other B-cell Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical College of Wisconsin (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065959; MCW-96110; MCW-HRRC-29196; NCI-V97-1368
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-10

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; Waldenström macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; primary systemic amyloidosis; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; sargramostim; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: cyclophosphamide
Drug: melphalan
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation in treating patients who have multiple myeloma or other B-cell cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of myeloablative therapy with autologous hematopoietic stem cell transplantation in patients with multiple myeloma and other B-cell malignancies.
* Determine the efficacy and pretransplantation prognostic factors associated with myeloablative therapy in these patients.
* Determine engraftment kinetics of granulocytes and platelets, as well as blood product transfusion requirements following hematopoietic stem cell transplantation.

OUTLINE: Patients must have hematopoietic stem cell procurement completed prior to myeloablative therapy. Patients receive high dose chemotherapy with autologous hematopoietic stem cell transplantation and supportive care. Melphalan is administered in one dose on day -1 at least 12 hours before stem cell infusion. Peripheral blood stem cells and/or bone marrow is reinfused on day 0. Filgrastim (G-CSF) or sargramostim (GM-CSF) is administered beginning on day 1 posttransplantation and continuing until blood counts recover.

Patients who are not candidates for tandem transplant may receive melphalan plus total body irradiation (TBI). Melphalan is administered IV on day -4. Total body irradiation is administered three times a day on days -3 and -2 and twice on day -1. At least 4 hours must elapse between each treatment. Hematopoietic stem cells are reinfused on day -1 upon completion of TBI or on day 0.

If patient is ineligible for melphalan plus TBI, the alternative single high dose regimen of melphalan plus cyclophosphamide is administered. Melphalan, for these patients, is given in two equal doses on day -4 followed by two consecutive days of cyclophosphamide on days -3 and -2. Hematopoietic stem cells are reinfused on day 0.

A second transplant may be considered, preferably between 3 and 6 months after the first transplant. The preferred regimen for the second transplant is melphalan alone or melphalan plus TBI as described above. The alternative regimens for the second dose therapy are melphalan alone or melphalan plus cyclophosphamide. For patients receiving melphalan alone, melphalan is administered in one dose on day -1 at least 12 hours before stem cell infusion. Hematopoietic stem cells are reinfused on day 0 for both alternative regimens.

Patients are followed for response from treatment for a minimum of 4 weeks and then periodically for survival.

PROJECTED ACCRUAL: A minimum of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma or other B-cell malignancy including non-Hodgkin's lymphoma, Waldenstrom's macroglobulinemia, or amyloidosis

  * Non-Hodgkin's lymphoma with T-cell immunophenotypes included

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3 (unless due to disease)
* Platelet count at least 100,000/mm^3 (unless due to disease)

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* LVEF at least 40%

Pulmonary:

* DLCO or FVC and FEV1 at least 50% of predicted unless due to restriction from volume loss secondary to disease

Other:

* HIV negative
* No overt infection or unexplained fever requiring broad spectrum antibiotics
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior biologic therapy

Chemotherapy:

* At least 2 weeks since other prior chemotherapy and recovered

Endocrine therapy:

* At least 2 weeks since prior endocrine therapy
* Concurrent steroids allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 1997-09

CONTACTS AND LOCATIONS:
Overall Officials: David H. Vesole, MD, PhD, Study Chair — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States